CLINICAL TRIAL: NCT00795548
Title: Phase-II Trial to Assess the Efficacy and Toxicity of 5-Azacitidine in Addition to Standard DLI for the Treatment of Patients With AML or MDS Relapsing After Allogeneic Stem Cell Transplantation
Brief Title: Safety Study of 5-Azacitidine and Standard Donor Lymphocyte Infusion (DLI) to Treat Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS) Relapsing After Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZARELA_HHU_2007
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: Myelodysplastic syndrome (MDS); Acute myeloid leukemia (AML); Stem cell transplantation; 5-Azacitidine; Donor lymphocyte infusion; MDS or AML relapsed after stem cell transplantation
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-Azacitidine (Experimental): 5-Azacitidine in addition to standard donor lymphocyte infusions.
  Interventions: Drug: 5-Azacitidine

INTERVENTIONS:
Drug: 5-Azacitidine — 5-Aza will be administered at doses of 100mg/m2 via subcutaneous injection over a period of 5 days. The total amount per treatment cycle, consisting of 5 days, is 500mg/m². Each treatment cycle is repeated every 28 days, with a treatment pause of 23 days between each 5-Aza cycle, to a total of 6 (optional 8 cycles) cycles.
  DLI will be transfused on day +34 with a total count of CD3+ cells of DLI 1-5x10E6CD3+/kg bodyweight. In absence of GvHD DLI transfusion is repeated on day +90 with DLI 1-5x10E7CD3+/kg bodyweight and on day +142 with DLI 1-5x10E8CD3+/kg bodyweight. Additional DLI may be given.
  Other Names: Vidaza

SUMMARY:
This open label phase-II trial evaluates hematological response of an additional treatment with 5-Azacitidine to common DLI in patients with MDS or AML relapsing after allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
Relapse after allogeneic stem cell transplantation is a major problem in patients with poor prognosis AML or MDS. Donor lymphocyte infusions alone re-induce remission in a minority of these patients, which may be the result of poor differentiation of the leukemic cells. The study drug 5-Aza is effective in AML and MDS.In addition to direct cytotoxicity, it alters gene expression and induces differentiation of leukemic blast cells. Furthermore, DNA-demethylating treatment results in an induction of transcription and cell surface expression of formerly unexpressed KIRs (killer Ig-like receptors) in NK cells, which are involved in the specific recognition of leukemic target cells and who are able to generate a specific graft-versus leukemia effect. The increased expression of MHC class I and II molecules on the surface of the recipient's leukemic cells and the de novo expression of formerly silenced KIR genes in donor NK cells due to treatment with 5-Aza may result in an increased susceptibility of myeloid leukemic cells to the allogeneic graft versus leukemia effect. Therefore, the graft-versus leukemia effect by donor lymphocyte infusions and NK cells from the original donor may be supported by additional therapy with 5-Azacitidine.

ELIGIBILITY:
Inclusion Criteria:

- Primary and secondary MDS, AML after MDS, and de novo AML relapsing after allogeneic stem cell transplantation

* Eligibility for Donor Lymphocyte Infusions
* Performance status according to the WHO scale: 0, 1 or 2.
* Adequate renal and liver function: bilirubin < 1.5 times the upper limit of normal and a GFR > 50 ml/min
* Absence of severe cardiovascular disease, i.e., arrhythmias requiring chronic treatment, congestive heart failure (NYHA Class III or IV) or symptomatic ischemic heart disease, where New-York Heart Association (NYHA)
* HIV negative and HBs-Ag negative.
* Absence of active uncontrolled infection (Septicaemia).
* No prior history or current evidence of central nervous system and psychiatric disorders requiring hospitalization.
* Age at least 18 years.
* Negative pregnancy test for women with reproductive potential.
* Signed written informed consent must be given according to national/local regulations.

Exclusion Criteria:

- Have malignant hepatic tumors.

* Severe liver dysfunction CHILD B and C.
* Renal insufficiency with a GFR < 50 ml/min
* Radiation therapy, chemotherapy, or cytotoxic therapy, given to treat conditions other than MDS, AML or applied for conditioning prior allogeneic stemcell transplantation.
* Psychiatric illness that would prevent granting of informed consent.
* Treatment with androgenic hormones during the previous 14 days prior Day 1.
* Active viral infection with known human immunodeficiency virus (HIV) or viral Hepatitis B or C.
* Hypersensitivity to Mannitol or 5-Azacitidine.
* Treatment with other investigational drugs following relapse after allogeneic stemcell transplantation or ongoing adverse events from previous treatment with investigational drugs regardless of time period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Best response | within the 6 months of treatment

SECONDARY OUTCOMES:
Safety and Toxicity of 5-Azacitidine for patients relapsing after allo-SCT | within 3 years
Response rate | within 6 months
Duration of remissions | within 3 years
Incidence of acute and chronic GvHD | 3 years
Achievement of complete chimerism | 6 month
Toxicity | wtihin 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guido Kobbe, PD Dr., Principal Investigator — Department of Hematology, Oncology and Clinical Immunology
Locations (6):
- Germany (6):
  - Universitaetsklinik Heidelberg, Medizinische Klinik und Poliklinik V, Heidelberg, Baden-Wurttemberg
  - Bone Marrow Transplantation Unit, University Hospital Hamburg-Eppendorf, Hamburg, Hamburg
  - Klinikum der Johann-Wolfgang-Goethe Universität, Medizinische Klinik II, Frankfurt am Main, Hesse
  - Department of Hematology, Oncology and Clinical Immunology, University Hospital Duesseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Dresden, Medizinische Klinik und Poliklinik I, Dresden, Saxony
  - Charite´-Campus Benjamin Franklin, Medizinische Klinik III, Berlin, State of Berlin